CLINICAL TRIAL: NCT05921071
Title: Do Patients Who Are Treated With Tranexamic Acid Loose Les Blood, Comparing to Patients Who Are Not Treated, During Vaginal Hysterectomy? a Randomized Control Study
Brief Title: Do Patients Who Received Tranexamic Acid in Vaginal Hysterectomy Loose Les Blood, Comparing to Patients Who Did Not?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Ohad Gluck, Senior gynecologist, Principal Investigator, Associated Professor, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: WOMC-22-0200
Record Dates: First submitted 2023-03-20; First posted 2023-06-27 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Vaginal Hysterectomy
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Randomized control
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic acid arm (Active Comparator): One gram of tranexamic acid (Hexakapron) is administered intravenously before surgery.
  Interventions: Drug: Tranexamic acid
- Placebo arm (Placebo Comparator): patients will receive 10 ml of normal saline 0.9% intravenously.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic acid — One gram of tranexamic acid (Hexakapron) is administered intravenously before surgery
  Other Names: Hexakapron
  Arms: Tranexamic acid arm
Drug: Placebo — patients will receive 10 ml of normal saline 0.9% intravenously.
  Other Names: Normal Selaine 0.9%
  Arms: Placebo arm

SUMMARY:
This is a randomized control, double-blind study in which women who are about to go an elective vaginal hysterectomy are offered to participate.

Patients will be randomly assigned to one of two groups: the tranexamic acid group, in which 1 gram of tranexamic acid (Hexakapron) is administered intravenously before surgery, and the control group, in which patients will receive 10 ml of normal saline 0.9% intravenously.

DETAILED DESCRIPTION:
This is a randomized control, double-blind study in which women who are about to go for an elective vaginal hysterectomy are offered to participate.

Patients will be randomly assigned to one of two groups: the tranexamic acid group, in which 1 gram of tranexamic acid (Hexakapron) is administered intravenously before surgery, and the control group, in which patients will receive 10 ml of normal saline 0.9% intravenously.

A nurse will prepare the solution according to the randomization and will handle it to the anesthesiologist.

ELIGIBILITY:
Inclusion Criteria:

*Women in general good health (defined as American Society of Anesthesiologists grade 1-2) who are about to undergo elective vaginal hysterectomy indicated by pelvic organ prolapse (POP).

Exclusion Criteria:

* allergy to TXA
* familial or personal history of hypercoagulability disorder or thromboembolic events
* impaired renal function or hematuria
* patients receiving antithrombotic therapy
* additional concurrent abdominal/ laparoscopic procedures
* malignancy
* Post-assignment exclusion will be executed in cases of conversion to laparotomy/ laparoscopy.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — only women
Enrollment: 80 (Estimated)
Dates: Start 2023-01-22 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Mean objective assessment of blood loss | Immediately after surgery
  Objective assessment of blood loss is calculated by subtraction the weight of used pads after the surgery from the preoperative weight (blood lost during surgery will be absorbed by pads only, without using suction); 1 g of absorbed fluid will be converted to 1 mL of blood.

SECONDARY OUTCOMES:
Mean subjective blood loss (SBL) | Immediately after surgery
  SBL will be estimated by the senior surgeon.
Mean difference in hemoglobin levels before and after surgery | One day after surgery
  Preoperative and postoperative hemoglobin level difference
The number of patients who need blood products transfusion | 30 days after surgery
  The need of blood transfusion or other blood products in order to treat excessive blood loss
The size of pelvic hematoma after surgery | One day after surgery
  Postoperative pelvic hematoma, diagnosed and measured by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Ohad Gluck, Principal Investigator — Wolfson Medical Center
Locations (1):
- Wolfson medical center, Holon, Israel